CLINICAL TRIAL: NCT00021398
Title: Phase II Study: Hyperfractionated Pre-Op Chemo-Radiation for Locally Advanced Rectal Cancer
Brief Title: Radiation Therapy and Chemotherapy Followed by Surgery and Combination Chemotherapy in Treating Patients With Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068776; P30CA006927 (NIH); FCCC-96071; NCI-G01-1988
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation Therapy, Chemotherapy and Surgery (Experimental)
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy and chemotherapy may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy and chemotherapy followed by surgery and combination chemotherapy in treating patients who have stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the local recurrence rate, disease-free survival, and overall survival of patients with stage II or III rectal cancer treated with neoadjuvant radiotherapy and fluorouracil followed by surgical resection and adjuvant fluorouracil and leucovorin calcium. II. Determine the toxicity rate in patients treated with this regimen. III. Correlate failure-free survival with ultrasound-determined preoperative staging in patients treated with this regimen. IV. Determine the quality of life of patients treated with this regimen. V. Determine if toxicity due to treatment, daily stool frequency, sexual dysfunction, and disease-free survival correlates with quality of life parameters in patients treated with this regimen. VI. Correlate clinical selection criteria with ability to perform sphincter-sparing surgery in patients treated with this regimen. VII. Determine post-chemoradiotherapy pathological response, margin status, and lymph node status and correlate these factors with initial clinico-pathologic findings in patients treated with this regimen.

OUTLINE: Patients undergo pelvic radiotherapy once daily five days a week for 5 weeks followed by boost radiotherapy twice daily for 7 days. Patients also receive neoadjuvant fluorouracil IV continuously over days 1-4 and 36-40. Patients undergo surgical resection 4-6 weeks after completion of radiotherapy. At 4 weeks after surgery, patients receive adjuvant leucovorin calcium IV and fluorouracil IV once daily five days a week. Treatment continues every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, at the completion of pelvic and boost radiotherapy, at 4 weeks after completion of chemoradiotherapy (prior to surgery), and then at 3, 6, and 12 months after completion of study therapy. Patients are followed every 3 months for 2 years, every 4 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 23-41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum
* Tumor extending through bowel wall (T3) OR
* Fixation to surrounding structures (T4) OR
* Nodal involvement by endorectal ultrasound (N1-2)
* Tumor extending through bowel wall, but not fixed (T3) must be:

  * At least 4 cm or at least 40% of bowel circumference OR
  * Accompanied by nodal involvement
* Evidence of transmural penetration confirmed by 2 of the following:

  * CT scan
  * Pelvic MRI
  * Transrectal ultrasound
  * Physical exam
* Proximal extent of tumor must not extend higher than 12 cm above dentate line and must be below pelvic peritoneal reflexion or sacral promontory
* Regional lymph node involvement allowed
* No distant metastases by CT scan of abdomen and pelvis or chest x-ray

PATIENT CHARACTERISTICS:

* Age: Over 18
* Performance status: ECOG 0-1
* Life expectancy: At least 2 years
* Hematopoietic:

  * Leukocyte count greater than 4,000/mm3
  * Platelet count at least 100,000/mm3
  * Hemoglobin greater than 10 g/dL
* Hepatic:

  * SGOT and SGPT less than 1.5 times normal
  * Bilirubin less than 1.5 mg/dL
* Renal: Creatinine less than 1.8 mg/dL
* Other:

  * Not pregnant or nursing
  * Negative pregnancy test
  * No other prior or concurrent malignancy within the past 5 years except inactive non-melanoma skin cancer or carcinoma in situ of the cervix
  * No psychiatric condition that would preclude informed consent
  * No other serious medical illness that would limit survival

PRIOR CONCURRENT THERAPY:

* Biologic therapy: Not specified
* Chemotherapy: No prior chemotherapy for rectal cancer
* Endocrine therapy: Not specified
* Radiotherapy: No prior radiotherapy for rectal cancer
* Surgery: No prior surgery for rectal cancer, except diagnostic biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1996-07; Primary Completion 2001-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Frequency of toxicity | weekly during treatment
tolerated dose of preoperative hyperfractionated radiation and concurrent chemotherapy | during radiation therapy and chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (17):
- United States (17):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Southern Chester County Medical Center, West Grove, Pennsylvania